CLINICAL TRIAL: NCT00047320
Title: A Phase II Study To Assess The Ability Of Neoadjuvant Chemotherapy Plus/Minus Second Look Surgery To Eliminate All Measurable Disease Prior To Radiotherapy For NGGCT
Brief Title: Neoadjuvant Chemotherapy With or Without Second-Look Surgery Followed by Radiation Therapy With or Without Peripheral Stem Cell Transplantation in Treating Patients With Intracranial Germ Cell Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0122; CDR0000257664 (Other: Clinical Trials.gov); COG-ACNS0122 (Other: Children's Oncology Group)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Brain Tumor; Central Nervous System Tumors; Childhood Germ Cell Tumor
Keywords: childhood central nervous system germ cell tumor; childhood teratoma; recurrent childhood malignant germ cell tumor; childhood central nervous system choriocarcinoma; childhood central nervous system embryonal tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor; recurrent childhood central nervous system embryonal tumor
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms; Teratoma | interventions — Carboplatin; Etoposide; etoposide phosphate; Ifosfamide; Thiotepa; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Peripheral Blood Stem Cell Transplantation; Radiotherapy; Craniospinal Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Therapy (CR from Induction) (Experimental): Patients will receive 6 cycles of Induction chemotherapy consisting of carboplatin and etoposide (Cycles 1, 3, and 5) alternating with ifosfamide and etoposide (Cycles 2, 4, and 6). The entire length of Induction is 18 weeks unless delay occurs due to myelosuppression or unanticipated toxicity. Each cycle of Induction will begin when ANC > 750/L and platelets > 75,000/L and when off filgrastim (G-CSF) for at least 48 hours. Following the Induction phase (weeks 0-18) those patient in CR will undergo radiation therapy.
  Interventions: Drug: carboplatin; Drug: etoposide; Drug: ifosfamide; Drug: thiotepa; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Given IV
  Other Names: Paraplatin; NSC #241240
Drug: etoposide — Given IV
  Other Names: VP-16; VePesid; Etopophos; NSC #141540
Drug: ifosfamide — Given IV
  Other Names: Isophosphamide; Iphosphamide; Z4942; Ifex; NSC #109724
Drug: thiotepa — Given IV
  Other Names: Tespa; Thiophosphamide; Triethylenethiophosphoramide Tspa; WR-45312; NSC #6396
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy — craniospinal irradiation
  Other Names: Craniospinal irradiation (CSI) followed by boost radiation to the sites of gross disease at diagnosis.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it is no longer present by conventional imaging and tumor markers from serum and cerebrospinal fluid. Radiation therapy uses high-energy x-rays to damage tumor cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Combining different types of therapy may kill more tumor cells.

PURPOSE: This Phase II trial is studying how well neoadjuvant chemotherapy with or without surgery and with or without high dose chemotherapy and peripheral stem cell transplantation, can increase response rates prior to radiation therapy and increase progression free and overall surviving patients with newly diagnosed intracranial germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with non-germinomatous germ cell tumors treated with neoadjuvant chemotherapy.
* Determine the progression-free survival and overall survival of patients treated with neoadjuvant chemotherapy with or without second-look surgery followed by radiotherapy with or without autologous peripheral blood stem cell transplantation (PBSCT).
* Determine whether additional complete responses can be achieved after high-dose thiotepa and etoposide with PBSCT in patients with persistently positive markers, histological evidence of residual malignant elements, or unresectable residual tumors after initial neoadjuvant chemotherapy.
* Determine patterns of recurrence in patients treated with this regimen.
* Correlate tumor marker response with radiographic and clinical measures of response, as well as findings at second-look surgery in patients with radiological evidence of residual disease.

OUTLINE:

* Induction chemotherapy:

  * Courses 1, 3, and 5: Patients receive carboplatin IV over 1 hour on day 1 and etoposide IV over 1 hour on days 1-3. Beginning on day 4, patients receive filgrastim (G-CSF) IV or subcutaneously (SC) for 10 days or until blood counts recover. Courses are 3 weeks in duration.
  * Courses 2, 4, and 6: Patients receive etoposide IV over 1 hour followed by ifosfamide IV over 1 hour on days 1-5. Beginning on day 6, patients receive G-CSF IV or SC for 10 days or until blood counts recover. Courses are 3 weeks in duration.

Patients undergo re-evaluation. Patients with a complete response (CR) go directly to radiotherapy. Approximately 3 weeks after completion of induction chemotherapy, all patients with less than a CR are encouraged to undergo second-look surgery.

After second-look surgery, patients with a CR or a partial response (PR) go directly to radiotherapy. Patients with less than a PR undergo consolidation chemotherapy with peripheral blood stem cell rescue (PBSC) followed by radiotherapy.

* Consolidation chemotherapy: Patients undergo PBSC collection. Patients receive G-CSF SC until PBSC collection is complete. Patients then receive thiotepa IV over 3 hours followed by etoposide IV over 3 hours on days -5 to -3. PBSCs are reinfused on day 0. Beginning on day 1 and continuing until blood counts recover, patients receive G-CSF SC daily.
* Radiotherapy: All patients receive radiotherapy once daily 5 days a week for 5-6 weeks beginning after recovery from induction chemotherapy or second-look surgery or within 9 weeks after PBSC reinfusion.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 80-100 patients will be accrued for this study within 36-42 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed intracranial non-germinomatous germ cell tumor (NGGCT) of 1 of the following types:

    * Endodermal sinus tumor (yolk sac tumor)
    * Embryonal carcinoma
    * Choriocarcinoma
    * Immature teratoma and teratoma with malignant transformation
    * Mixed germ cell tumor
  * Histologically confirmed germinoma with elevation of serum/CSF beta human chorionic gonadotropin (HCG) levels greater than 50 mIU/mL or any serum/CSF alpha-fetoprotein (AFP) levels greater than 10 ng/ml or above institutional norm
  * Histologically unconfirmed pineal and/or suprasellar tumors with serum/CSF beta HCG levels greater than 50 mIU/mL or AFP levels greater than 10 ng/ml or above institutional norm
* Patients with normal AFP and beta HCG < 50 mIU/mL without histologic diagnosis of a NGGCT or patients with pure germinoma without elevation of tumor marker are ineligible
* Initial diagnosis within the past 31 days

PATIENT CHARACTERISTICS:

Age

* 3 to 24 at diagnosis

Performance status

* No minimum performance level

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 10.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Pulmonary

* No assisted ventilation

Other

* Seizure disorders allowed
* No patients in status or coma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patient must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Prior corticosteroids allowed
* Concurrent corticosteroids allowed
* Concurrent endocrine replacement therapy allowed (e.g., L-thyroxine, testosterone, estrogen, desmopressin acetate)
* No concurrent growth hormone therapy

Radiotherapy

* Not specified

Surgery

* More than 1 prior surgery allowed

Other

* No other prior therapy for malignancy

Ages: 3 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2004-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, MD, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (106):
- United States (90):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (9):
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (2):
  - Starship Children's Health, Auckland
  - Christchurch Hospital, Christchurch
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva

REFERENCES:
- [Derived] Fangusaro J, Wu S, MacDonald S, Murphy E, Shaw D, Bartels U, Khatua S, Souweidane M, Lu HM, Morris D, Panigrahy A, Onar-Thomas A, Fouladi M, Gajjar A, Dhall G. Phase II Trial of Response-Based Radiation Therapy for Patients With Localized CNS Nongerminomatous Germ Cell Tumors: A Children's Oncology Group Study. J Clin Oncol. 2019 Dec 1;37(34):3283-3290. doi: 10.1200/JCO.19.00701. Epub 2019 Sep 23. PMID 31545689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy (CR From Induction)
Started | 104
Completed | 76
Not Completed | 28
Not completed — Lack of Efficacy | 8
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 8
Not completed — Withdrawal by Subject | 9
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 104
Age, Continuous [Median (Full Range); unit: years] | 12 [3 to 23]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 9
  White | 72
  More than one race | 0
  Unknown or Not Reported | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 85
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 88
  Canada | 10
  Australia | 5
  New Zealand | 1

OUTCOME MEASURES:

1. Primary Outcome: Response to Induction Chemotherapy
Description: A patient who achieves a complete or partial response, defined a reduction of at least 65% in tumor size after induction chemotherapy will be considered to have experienced response.
Time Frame: 18 weeks
Population: Of the 102 eligible patients, 85 completed induction chemotherapy with sufficient data to assess response. Central review response assessment is used.
Measure: Count of Participants; unit: Participants
Groups:
- Radiation Therapy (CR From Induction): Patients will receive 6 cycles of Induction chemotherapy consisting of carboplatin and etoposide (Cycles 1, 3, and 5) alternating with ifosfamide and etoposide (Cycles 2, 4, and 6). The entire length of Induction is 18 weeks unless delay occurs due to myelosuppression or unanticipated toxicity. Each cycle of Induction will begin when ANC > 750/L and platelets > 75,000/L and when off filgrastim (G-CSF) for at least 48 hours. Following the Induction phase (weeks 0-18) those patient in CR will undergo radiation therapy.
  carboplatin: Given IV
  etoposide: Given IV
  ifosfamide: Given IV
  thiotepa: Given IV
  adjuvant therapy
  conventional surgery
  neoadjuvant therapy
  peripheral blood stem cell transplantation
  radiation therapy: craniospinal irradiation
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 85
Participants
  Responder | 74
  Non-Responder | 11

2. Secondary Outcome: The Probability of Event-free Survival (EFS)
Description: Event-free Survival was defined as time from study entry to death from any cause, disease progression or recurrence, or second malignant neoplasm. Event-free survival was estimated by KM estimate.
Time Frame: At 3 years from study entry
Population: Two ineligible patients were excluded. A total of 102 eligible patients were analyzed.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 102
Probability | 0.837 [0.763 to 0.910]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free Survival was defined as time from study entry to disease progression or recurrence. Deaths that are clearly unrelated to disease progression, and second neoplasms are censored in this analysis. Progression -free survival was estimated by KM estimate.
Time Frame: At 3 years from study entry
Population: Two ineligible patients were excluded. A total of 102 eligible patients were analyzed. one patient died without the disease progression reported. But the death was due to the disease. The death was counted as "event" when progression-free survival (PFS) was calculated. So EFS and PFS at 3 years were same.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 102
Probability | 0.837 [0.763 to 0.910]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival was defined as time from study entry to death from any cause. Overall survival was estimated by KM estimate.
Time Frame: At 3 years from study entry
Population: Two ineligible patients were excluded. A total of 102 eligible patients were analyzed.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 102
Probability | 0.927 [0.876 to 0.979]

5. Secondary Outcome: Number of Patients Experiencing Toxic Death
Description: Toxic death, defined as death predominantly attributable to treatment-related causes.
Time Frame: During chemotherapy (up to 18 weeks)
Population: A total of 102 eligible patients treated with induction chemotherapy were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 102
Participants | 0

6. Secondary Outcome: Occurrence of Non-hematological Grade 4 Toxicity Occurrence of Nonhematological Grade 4 Toxicity
Description: The number of patients who experienced non-hematological grade 4 toxicities anytime during chemotherapy.
Time Frame: During chemotherapy(up to 18 weeks)
Population: A total of 102 eligible patients treated with induction chemotherapy were included.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Radiation Therapy (CR From Induction)
Number analyzed (Participants) | 102
participants | 22 [14 to 31]

ADVERSE EVENTS:
Description: 104 patients enrolled, 2 are ineligible and not included in adverse event reporting. Therefore, adverse events participants reported is 102.
Arm/Group | Radiation Therapy (CR From Induction)
Serious Adverse Events (participants affected / at risk) | 8/102
Other Adverse Events (participants affected / at risk) | 70/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (CR From Induction) (N=102)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (CR From Induction) (N=102)
Anemia (Blood and lymphatic system disorders) | 51 (108)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9)
Nausea (Gastrointestinal disorders) | 8 (16)
Vomiting (Gastrointestinal disorders) | 15 (28)
Infections and infestations - Other, specify (Infections and infestations) | 8 (10)
Alanine aminotransferase increased (Investigations) | 23 (39)
Aspartate aminotransferase increased (Investigations) | 15 (22)
Lymphocyte count decreased (Investigations) | 19 (42)
Neutrophil count decreased (Investigations) | 53 (104)
Platelet count decreased (Investigations) | 53 (96)
White blood cell decreased (Investigations) | 48 (114)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (37)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 10 (11)
Hypernatremia (Metabolism and nutrition disorders) | 20 (32)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 15 (22)
Hypokalemia (Metabolism and nutrition disorders) | 26 (39)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (13)
Hyponatremia (Metabolism and nutrition disorders) | 31 (57)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (12)
Headache (Nervous system disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.